CLINICAL TRIAL: NCT07173036
Title: Evaluation of (Cardio)Metabolic and Auxological Outcomes of GHD Patients Under Recombinant Human or Long-acting Growth Hormone With Stratification According to IGF-1 Levels
Brief Title: Evaluation of (Cardio)Metabolic and Auxological Outcomes of GHD Patients Under rhGH or LAGH With Stratification According to IGF-1 Levels
Acronym: METAB-BELGROW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/02JUI/216
Record Dates: First submitted 2025-06-13; First posted 2025-09-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Growth Hormone Deficiency
Keywords: metabolic outcomes; auxological outcomes; recombinant human growth hormone; long acting growth hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Metabolic Networks and Pathways

STUDY DESIGN:
Intervention Model Description: Patients will be classified into two groups (depending on their treatment as decided by their pediatric endocrinologist):
  * patients with GHD who receive daily rhGH= rhGH cohort
  * patients with GHD who receive weekly LAGH= LAGH cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhGH cohort (Other): Patients with GHD who receive daily rhGH (dose titration according to guidelines i.e. 25-35 micrograms/kg body weight/day)
  Interventions: Other: metabolic and auxological outcomes
- LAGH cohort (Other): Patients with GHD who receive weekly LAGH (dose titration according to guidelines i.e. for somatrogon 0.66 milligrams/kg body weight/week)
  Interventions: Other: metabolic and auxological outcomes

INTERVENTIONS:
Other: metabolic and auxological outcomes — Evaluation over a three-year period following the initiation of treatment with daily recombinant human growth hormone (rhGH)
  Arms: rhGH cohort
Other: metabolic and auxological outcomes — Evaluation over a three-year period following the initiation of treatment with weekly long-acting growth hormone (LAGH).
  Arms: LAGH cohort

SUMMARY:
The METAB-BELGROW-LAGH study aims to prospectively evaluate the metabolic outcomes of Belgian children diagnosed with growth hormone deficiency (GHD) over a three-year period following the initiation of treatment with either daily recombinant human growth hormone (rhGH) or weekly long-acting growth hormone (LAGH). Patients will be stratified according to their IGF-1 levels. The primary objective is to assess the metabolic outcomes of children treated with daily rhGH over the first three years. The secondary objectives include comparing the metabolic outcomes between patients treated with daily rhGH and those treated with weekly LAGH, and characterizing metabolic profiles based on IGF-1 levels. To achieve these objectives, both standard-of-care (SOC) and additional data will be collected at scheduled follow-up visits (baseline, 6, 12, 24, and 36 months), including clinical, auxological, and biological parameters. Additional metabolic markers, inflammatory and endothelial biomarkers will be assessed. In a subset of patients, carotid intima-media thickness (cIMT) and body fat distribution (via DEXA-scan) will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with growth hormone deficiency (GHD)
* Treated with growth hormone (rhGH or LAGH)

Exclusion Criteria:

* No exclusion criteria

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Auxological evaluation_1 | 3 years
  Primary outcome measures included change in stature (in cm and SDS) over the course of the study.
Auxological evaluation_2 | 3 years
  Primary outcome measures included change in weight (in kgs and SDS) over the course of the study.
Auxological evaluation_3 | 3 years
  Primary outcome measures included change in BMI (in kg/m2) over the course of the study.
Evaluation of the blood pressure | 3 years
  Measure of the systolic and diastolic blood pressure (in mmHg) with a sphygmomanometer
Evaluation of waist circumference | 3 years
  Measure of waist circumference (in cm) with a meter
Evaluation of clinical signs of puberty (Tanner stage) and androgenism | 3 years
  Evaluation of clinical signs of puberty (Tanner stage) and androgenism.
Metabolic evaluation_1 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of fasting glycemia (mg/dl).
Metabolic evaluation_2 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of fasting insulin (pmol/L).
Metabolic evaluation_3 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of hemoglobin A1c in diabetic patients (%).
Metabolic evaluation_4 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of transaminases (UI/L).
Metabolic evaluation_5 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of lipid profile (mg/dL).
Metabolic evaluation_6 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of creatinine (mg/dL).
Metabolic evaluation_7 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of alkaline phosphatase (UI/L).
Metabolic evaluation_8 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of calcium (mmol/L).
Metabolic evaluation_9 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of phosphorus (mmol/L).
Metabolic evaluation_10 | 3 years
  Evaluation of the change of the metabolic profile using both SOC and non-SOC Blood tests samples. Measurements of insulin-like growth factor 1 levels (ng/mL).
Bone markers_1 | 3 years
  Measurements in blood samples of bone markers such as procollagen type 1 N-terminal propeptide (µg/L).
Bone markers_2 | 3 years
  Measurements in blood samples of bone markers such as insulin-like growth factor (ng/mL).
Bone markers_3 | 3 years
  Measurements in blood samples of bone markers such as insulin-like growth factor binding protein (µL/mL).
Endothelial stress and inflammatory markers_1 | 3 years
  Measurements in blood samples of endothelial stress and inflammatory markers such as asymmetric dimethylarginine (µmol/L).
Endothelial stress and inflammatory markers_2 | 3 years
  Measurements in blood samples of endothelial stress and inflammatory markers such as TNF-a (pg/mL).
Endothelial stress and inflammatory markers_3 | 3 years
  Measurements in blood samples of endothelial stress and inflammatory markers such as VEGF (pg/mL).
Endothelial stress and inflammatory markers_4 | 3 years
  Measurements in blood samples of endothelial stress and inflammatory markers such as IL-6 (pg/mL).
Radiological evaluation of cIMT | 3 years
  Measurements of cIMT (mm) using Doppler ultrasound.
Radiological evaluation of body fat distribution | 3 years
  Measurements of body fat distribution (g/cm2) using DEXA-Scan.

SECONDARY OUTCOMES:
comparison with patients under weekly LAGH | 3 years
  Data obtained for patients with daily rhGH will be compared to data obtained for patients with weekly LAGH treatment.
  Same measurement description as for the primary outcomes.
Stratification of the metabolic profile of the patients according to IGF-1 levels | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lysy, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No